CLINICAL TRIAL: NCT01752309
Title: The Predictive Value of Ultrasound in Early Rheumatoid Arthritis
Acronym: EVA
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Maasstad Hospital (Other); Albert Schweitzer Hospital (Other); Vlietland Ziekenhuis (Other); UMC Utrecht (Other); Medical Center Alkmaar (Other); Ziekenhuisgroep Twente (Other)
Responsible Party: Principal Investigator, Ten Cate, David F. Ten Cate, MD, Erasmus Medical Center
Other Study IDs: MEC2009-333; NL28038.078.09 (Registry Identifier: CCMO)
Record Dates: First submitted 2012-12-12; First posted 2012-12-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Rheumatoid Arthritis; Predictive Value of Ultrasound in Early Rheumatoid Arthritis
Keywords: Early Rheumatoid arthritis; Rheumatoid arthritis; Ultrasound; Predictive; Prognosis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rheumatoid Arthritis, ultrasound, persistence disease activity: Patients diagnosed with early Rheumatoid Arthritis will be assessed three times in one year with ultrasound to evaluate the predictive value of ultrasound.

SUMMARY:
Rheumatoid arthritis a chronic and progressive inflammatory disease characterized by synovial membrane inflammation, possibly leading to destruction of joints. To start early with a combination therapy results in a better outcome for patients. Using ultrasonography it is possible to detect clinically and radiographically absent synovitis and erosions. However, it is unclear whether or not these findings have predictive value in these patients regarding disease activity or radiographical progression.

DETAILED DESCRIPTION:
Patients will be evaluated using the standard diagnostic workup of patients with early arthritis. This includes history taking, physical examination, Disease Activity Score of 44 joints (DAS44) and a laboratory test, including C-Reactive Protein(CRP), Erythrocyte Sedimentation Rate (ESR), Complete Blood Count (CBC), Rheumatoid Factor (RF), Anti-Cyclic Citrullinated Peptide(anti-CCP), transaminases, urinanalysis.

Also part of the standard workup for these patients are X-Rays of hands and feet to detect erosions. The baseline medication will include - in concordance with European League Against Rheumatism (EULAR)-guidelines and the provisional 'Nederlandse Vereniging voor Reumatologie(NVR)'-guidelines - Methotrexate (MTX) for all patients. The medicine regimes are part of the ongoing cohort studies from which the patients will be recruited. Evaluating the medicine effects is not part of the 'Echografie bij Vroege Artritis (EVA)(Ultrasound in Early Arthritis)' study. All consecutive Rheumatoid Arthritis (RA) patients will be asked to participate in this study. They will receive oral and written information about the EVA study.

Approximately two weeks after this first consultation the patient returns to his or her rheumatologist for the diagnosis and accompanying treatment. If the patient decides to participate in this study they fill out the informed consent form. The patient will be asked to fill out the Health Assessment Questionnaire (HAQ) and the Short Form-36 (SF-36). After this, at baseline, at three months and at 12 months, Metatarsophalangeal (MTP) 2-5(dorsal aspect) and Metacarpophalangeal (MCP) 2-5(dorsal, palmar, lateral) and wrists of each patient will be examined with ultrasound by a single rheumatologist per centre specialized in Ultrasound (US). This rheumatologist will be unaware of the clinical, laboratory and radiographic findings.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed rheumatoid arthritis patients, diagnosed according to the American College of Rheumatology (ACR) 1987-criteria
* Naïve for Disease Modifying Anti Rheumatic Drugs (DMARDs), biologicals and glucocorticoids.
* Starting with treatment with a potent anti-rheumaticum. E.g. methotrexate (MTX), biologicals or glucocorticoids.

Exclusion Criteria:

* Contra-indications for MTX, biologicals or glucocorticoids.
* Insufficient ability to read and write in Dutch
* Personality disorders that limit the participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Starting in June 2010, all newly diagnosed rheumatoid arthritis patients who will be participating in 2 ongoing trials will be invited to participate in this study. In Almelo they will be recruited from the outpatient Rheumatology clinic.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Persistence of active disease after one year, defined as a Disease Activity Score of 44 joints (DAS44) > 3.4 | One year after inclusion in the study

SECONDARY OUTCOMES:
Change in Sharp vd Heijde score during the year of inclusion | At date of inclusion and after one year

OTHER OUTCOMES:
Change of DAS over time | At date of inclusion, after 3 months and after one year

CONTACTS AND LOCATIONS:
Overall Officials: Jolanda J. Luime, PhD, Principal Investigator — Erasmus Medical Center
Locations (7):
- Netherlands (7):
  - Medical Center Alkmaar, Alkmaar, North Holland
  - Ziekenhuisgroep Twente, Almelo, Overijssel
  - Albert Schweitzer Hospital, Dordrecht, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - Maasstad Hospital, Rotterdam, South Holland
  - Vlietland Hospital, Schiedam, South Holland
  - University Medical Center Utrecht, Utrecht, Utrecht

REFERENCES:
- [Derived] Ten Cate DF, Jacobs JWG, Swen WAA, Hazes JMW, de Jager MH, Basoski NM, Haagsma CJ, Luime JJ, Gerards AH. Can baseline ultrasound results help to predict failure to achieve DAS28 remission after 1 year of tight control treatment in early RA patients? Arthritis Res Ther. 2018 Jan 30;20(1):15. doi: 10.1186/s13075-018-1514-2. PMID 29382379